CLINICAL TRIAL: NCT06654063
Title: Clinical Assessment of Adjunctive Omega-3 Versus Vitamin D Daily Supplements on Active Periodontal Therapy With Stage II Grade B Periodontitis Patients: A Randomized Controlled Clinical Trial.
Brief Title: Clinical Assessment of Adjunctive Omega-3 Versus Vitamin D Daily Supplements on Active Periodontal Therapy With Stage II Grade B Periodontitis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Helal, Lecturer Periodontology and implantology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 531024
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non-surgical periodontal therapy (SRP) (Active Comparator): * The CAL PPD and mSBI will be measured for each patient and will be recorded at baseline and 6 weeks
  * all patients will receive supragingival and sub-gingival plaque and calculus debridement (SRP) with an ultrasonic scaler (Various 350; NSK, Japan) and a manual universal curette (Gracey; Hu-Friday, Chicago, USA) where, conventional scaling and root planning (SRP) to the bottom of the pocket of 4 mm or more
  * Subgingival saline irrigation will be performed adjunctively to Sub-gingival curettage.
  Interventions: Procedure: non-surgical periodontal therapy (SRP); Dietary Supplement: non-surgical periodontal therapy (SRP)+ Omega-3; Dietary Supplement: non-surgical periodontal therapy (SRP)+ Vitamin D
- non-surgical periodontal therapy (SRP)+ Omega-3 (Experimental): * The CAL PPD and mSBI will be measured for each patient and will be recorded at baseline and 6 weeks
  * patients will receive supragingival and sub-gingival plaque and calculus debridement (SRP) with an ultrasonic scaler (Various 350; NSK, Japan) and a manual universal curette (Gracey; Hu-Friday, Chicago, USA)
  * Subgingival saline irrigation will be performed adjunctively to Sub-gingival curettage.
  * Patients will start taking Omega-3 supplements on the day of SRP procedure.
  Interventions: Procedure: non-surgical periodontal therapy (SRP); Dietary Supplement: non-surgical periodontal therapy (SRP)+ Omega-3; Dietary Supplement: non-surgical periodontal therapy (SRP)+ Vitamin D
- non-surgical periodontal therapy (SRP)+ Vitamin D (Experimental): * Patients will start taking Omega-3 supplements on the day of SRP procedure.
  * Serum vitamin D levels will be assessed at baseline and 6 weeks after intervention in all groups.
  Interventions: Procedure: non-surgical periodontal therapy (SRP); Dietary Supplement: non-surgical periodontal therapy (SRP)+ Omega-3; Dietary Supplement: non-surgical periodontal therapy (SRP)+ Vitamin D

INTERVENTIONS:
Procedure: non-surgical periodontal therapy (SRP) — * The CAL PPD and mSBI will be measured for each patient and will be recorded at baseline and 6 weeks
  * all patients will receive supragingival and sub-gingival plaque and calculus debridement (SRP) with an ultrasonic scaler (Various 350; NSK, Japan) and a manual universal curette (Gracey; Hu-Friday, Chicago, USA) where, conventional scaling and root planning (SRP) to the bottom of the pocket of 4 mm or more
  * Subgingival saline irrigation will be performed adjunctively to Sub-gingival curettage.
Dietary Supplement: non-surgical periodontal therapy (SRP)+ Omega-3 — * The CAL PPD and mSBI will be measured for each patient and will be recorded at baseline and 6 weeks
  * all patients will receive supragingival and sub-gingival plaque and calculus debridement (SRP) with an ultrasonic scaler (Various 350; NSK, Japan) and a manual universal curette (Gracey; Hu-Friday, Chicago, USA)
  * Subgingival saline irrigation will be performed adjunctively to Sub-gingival curettage.
  * Patients will start taking Omega-3 supplements on the day of SRP procedure.
Dietary Supplement: non-surgical periodontal therapy (SRP)+ Vitamin D — * The CAL PPD and mSBI will be measured for each patient and will be recorded at baseline and 6 weeks
  * all patients will receive supragingival and sub-gingival plaque and calculus debridement (SRP) with an ultrasonic scaler (Various 350; NSK, Japan) and a manual universal curette (Gracey; Hu-Friday, Chicago, USA) where, conventional scaling and root planning (SRP) to the bottom of the pocket of 4 mm or more
  * Subgingival saline irrigation will be performed adjunctively to Sub-gingival curettage.
  * Serum vitamin D levels will be assessed at baseline and 6 weeks after intervention in all groups.

SUMMARY:
Clinical Assessment of Adjunctive Omega-3 Versus Vitamin D daily Supplements on Active Periodontal Therapy with Stage II Grade B Periodontitis Patients: A Randomized controlled clinical trial.

DETAILED DESCRIPTION:
This randomized clinical trial evaluates the effect of Omega- 3 versus Vitamin D regarding Clinical evaluation

1. Clinical attachment loss (CAL)
2. Plaque index (PI)
3. Gingival index (GI)

ELIGIBILITY:
Inclusion Criteria:

* • Systemic healthy patients

  * Patients aged > 25 years
  * Patients suffering from stage II periodontitis with grade B were included in this study, according to 2017 world workshop classification of periodontal disease (Papapanou et al. 2017).
  * Patients with interdental clinical attachment loss (CAL) of 3-4 mm
  * No history of previous periodontal therapy.
  * No taken medications known to interfere healing or periodontal tissue health such as anticonvulsants, calcium channel blockers, or immunosuppressant drugs.
  * No previous periodontal surgery at involved sites.
  * Good oral hygiene and good compliance with the plaque control instructions following initial therapy.
  * Neither taken antibiotics within the last three months nor nonsteroidal anti-inflammatory drugs within the last three months
  * Absence of diseases or conditions that would interfere with wound healing such as diabetes mellitus or coagulation disorders
  * Absence of oral mucosal inflammatory conditions such as aphthous ulcers or lichen planus.

Exclusion Criteria:

* • Patients taking Omega- 3 or Vitamin D as a nutritional supplement were excluded from the study

  * Smoking habits
  * Pregnant and lactating mothers
  * Patients who have been received periodontal surgery in the study area during the last 6 months.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical attachment loss (CAL) | Day 0 - month 3- month 6
  * All clinical outcomes will be measured baseline, 6 weeks after SRP alone and in conjunction with Omega- 3 and Vitamin D.
  * CAL will be measured form cemento- enamel junction (CEJ) to the depth of the pocket using UNC periodontal probe.
  * It will be recorded at 6 sites per tooth, the recorded readings will be used to generate mean values at each time point.

SECONDARY OUTCOMES:
Plaque index (PI) | Day 0 - month 3- month 6
  • through the Silness & Loe plaque index score: score the thickness of plaque, sum the scores, and divide by the number of surfaces/teeth to get an average score. 0: no plaque - 1: thin film on gingival margin - 2: visible plaque in pocket and on gingival margin - 3: dense plaque in pocket and on gingival margin
Gingival index (GI) | Day 0- month 3- month 6
  through the modified Loe & Silness score by assigning a score to each site based on these criteria as follows. 0: normal gingiva - 2: mild inflammation (slight color change, slight edema, no bleeding on probing) - 3: moderate inflammation (redness-edema-glazing-bleeding on probing) - 3: severe inflammation (marked redness, edema, spontaneous bleeding, or ulceration).

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Helal, Cairo, Egypt